CLINICAL TRIAL: NCT05904860
Title: Effects of Backward vs Forward Gait Training With Auditory Feedback in Patients With Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shifa Tameer-e-Millat University (Other)
Responsible Party: Principal Investigator, Nouman Khan, Lecturer, Shifa Tameer-e-Millat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB 0350-22
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Stroke, Ischemic
Keywords: Stroke, Gait Training, Auditory feedback
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Intervention Model Description: total two groups are formed with 22 participants in each group. One is the treatment group which will receive backward gait training. The other is the control group receiving forward gait training. Pre-intervention outcomes are measured. Followed by mid-protocol outcome measurement after 2 weeks and end-protocol measurement after 4 weeks.
Who Masked: Participant
Masking Description: Participants of the study are not informed in which group they are placed. The placement of the group is selected through the sealed envelope method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Other): The experimental group will be receiving a 30-minute backward gait training using parallel bars, a mirror, and on a firm surface. Patients will receive training for 4 days per week with a total time period of 4 weeks. Balance, fall risk, and spatiotemporal gait parameters will be quantified and evaluated before the commencement of treatment, after 2 weeks, and at the end of the last session.
  Interventions: Other: Backward Gait Training
- Control group (Other): The control group will be receiving a 30-minute forward gait training using parallel bars, a mirror and on a firm surface. Patients will receive training for 4 days per week with a total time period of 4 weeks. Balance, fall risk, and spatiotemporal gait parameters will be quantified and evaluated before the commencement of treatment, after 2 weeks, and at the end of the last session.
  Interventions: Other: Forward Gait Training

INTERVENTIONS:
Other: Backward Gait Training — Backward gait training will be provided within parallel bars, a mirror, and on a firm surface. The harness belt will be around the patient's torso to avoid sudden falls.
  Other Names: Auditory Feedback
  Arms: Experimental Group
Other: Forward Gait Training — Forward gait training will be provided within parallel bars, a mirror, and on a firm surface. The harness belt will be around the patient's torso to avoid sudden falls.
  Other Names: Auditory Feedback
  Arms: Control group

SUMMARY:
One of the major expressions of chronic disability in patients with cerebrovascular accidents is in terms of impaired gait and balance. Both of these limitations have an ultimate effect in terms of increased risk of falls leading to augmented morbidity and mortality. Further results of gait abnormalities and balance impairments are increased morbidity with many other manifestations including but not limited to; pain, a significant reduction in quality of life, muscle as well as joint stiffness, postural instability self-imposed restricted physical functioning, and limited social interaction. The chances of an acute recurrent stroke are substantially increased due to restricted mobility.

DETAILED DESCRIPTION:
A variety of treatment options are available for balance improvement and gait training in stroke patients including conventional treatment options of stretching, muscle strengthening, limb stabilization joint mobilizations followed by forward walking training with or without support and modern technological advancements including virtual reality immersion exercises, motor imagery and hydro treadmill. However, backward walking, also known as retro gait, is the emerging key therapy for gait training. Neuronal circuits located inside the spinal cord and brainstem; known as central pattern generators (CPGs), are primarily responsible for producing automated outputs for rhythmic motor responses example ambulation. These CPGs, along with the descending system, are responsible for motor neuron activation by setting the threshold muscle lengths. The CPGs that are responsible for forward ambulation, also regulate the backward gait. A more intensified recruitment of lower limb musculature motor unit has been observed during backward gait in individuals. Also, due to the restricted visual field when walking backward, the temporal and spatial gait parameters are significantly increased. For the aforementioned reasons, backward gait training can be used as an alternative strategy to improve balance and ambulation.

The performance of an individual during motor relearning can be influenced by using a stimulus from an external source that will generate a behavioral response leading to self-modification in motor action known as a biofeedback system. The most common types of biofeedback include visual, auditory as well as tactile stimuli that inform the individual involved in biofeedback training, about his relative achievements in reaching gait and balance-related targets. Recent literature proposes the notion that in a comparison of visual biofeedback versus auditory biofeedback, individuals under study are more prone to develop a dependence on external cues when using visual biofeedback. Also, poor performance was demonstrated by individuals receiving training with visual feedback on motor retention tests as compared to the individuals receiving auditory feedback. Thus auditory feedback tends to be more helpful in terms of motor relearning.

Backward walking training activates the central pattern generators that are responsible for ambulation however, muscle fiber recruitment had been observed to be more intensified as compared to recruitment during forward gait training. Forward gait training with auditory biofeedback effectively improves stride length, balance, and walking speed in individuals with stroke.

Since backward gait training has a more pronounced effect on gait parameters as compared to forward walking, also, in the light of recent evidence motor re-learning can be enhanced using biofeedback, the combined effect of backward gait training with auditory biofeedback could produce more pronounced effects in terms of motor recovery and improved balance and decreased risk of fall as compared to conventional forward gait training with biofeedback.

ELIGIBILITY:
Inclusion Criteria:

Both genders First-time ischemic stroke Diagnosed Middle cerebral artery stroke patients Sub-acute stroke 3 weeks- 11 weeks Hemiplegia Age 35 years to 65 years Brunnstorm's stages 4 to 6 Able to maintain standing posture with minimum assistance with a Berg balance scale score greater than 45

Exclusion Criteria:

GCS lower than 15 Any other neurological diagnosis Presence of associated cognitive impairment Lower extremity joint deformities Any prominent visual problem hindering ambulation Patients with auditory compromise and patients using hearing aids

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-06-06 (Actual); Primary Completion 2023-07-11 (Estimated); Study Completion 2023-07-25 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale | 4 weeks
  It is a 14 items static and dynamic balance measurement tool. The total score on this scale is 56 with 4 maximum scores in each item. Higher scores demonstrate good balance. Lower scores demonstrate poor balance.
Cadence | 4 weeks
  Pedometers are designed to detect vertical movement at the hip and so measure the number of steps and provide an estimate of the distance walked. They cannot provide information on the temporal pattern of physical activity or the time spent in different activities at different intensities.
Walking Speed | 4 weeks
  walking speed that would be calculated using formula "Walking speed = distance covered / time taken
Stride Length | 4 weeks
  stride length that would be calculated using formula "Stride length = Distance covered / (1/2x cadence)
Step Length | 4 weeks
  step length that would be calculated using formula "Step length = stride length / 2

CONTACTS AND LOCATIONS:
Overall Officials: Noor-ul-ain Sohail, MS-PT*, Principal Investigator — Shifa Tameer-e-Millat University
Locations (1):
- Shifa Tameer-e-Millat University Islamabad, Islamabad, Fedral, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Balasukumaran T, Olivier B, Ntsiea MV. The effectiveness of backward walking as a treatment for people with gait impairments: a systematic review and meta-analysis. Clin Rehabil. 2019 Feb;33(2):171-182. doi: 10.1177/0269215518801430. Epub 2018 Sep 19. PMID 30229667
- [Background] Bytyci I, Henein MY. Stride Length Predicts Adverse Clinical Events in Older Adults: A Systematic Review and Meta-Analysis. J Clin Med. 2021 Jun 17;10(12):2670. doi: 10.3390/jcm10122670. PMID 34204430
- [Background] Cha YJ, Kim JD, Choi YR, Kim NH, Son SM. Effects of gait training with auditory feedback on walking and balancing ability in adults after hemiplegic stroke: a preliminary, randomized, controlled study. Int J Rehabil Res. 2018 Sep;41(3):239-243. doi: 10.1097/MRR.0000000000000295. PMID 29782407
- [Background] Feldman AG, Levin MF, Garofolini A, Piscitelli D, Zhang L. Central pattern generator and human locomotion in the context of referent control of motor actions. Clin Neurophysiol. 2021 Nov;132(11):2870-2889. doi: 10.1016/j.clinph.2021.08.016. Epub 2021 Sep 27. PMID 34628342
- [Background] Kondo K, Noonan KM, Freeman M, Ayers C, Morasco BJ, Kansagara D. Efficacy of Biofeedback for Medical Conditions: an Evidence Map. J Gen Intern Med. 2019 Dec;34(12):2883-2893. doi: 10.1007/s11606-019-05215-z. Epub 2019 Aug 14. PMID 31414354
- [Background] Maier M, Ballester BR, Verschure PFMJ. Principles of Neurorehabilitation After Stroke Based on Motor Learning and Brain Plasticity Mechanisms. Front Syst Neurosci. 2019 Dec 17;13:74. doi: 10.3389/fnsys.2019.00074. eCollection 2019. PMID 31920570
- [Background] McLellan AG, Slaght J, Craig CM, Mayo A, Senechal M, Bouchard DR. Can older adults improve the identification of moderate intensity using walking cadence? Aging Clin Exp Res. 2018 Jan;30(1):89-92. doi: 10.1007/s40520-017-0746-3. Epub 2017 Apr 4. PMID 28378230
- [Background] Park C, Oh-Park M, Dohle C, Bialek A, Friel K, Edwards D, Krebs HI, You JSH. Effects of innovative hip-knee-ankle interlimb coordinated robot training on ambulation, cardiopulmonary function, depression, and fall confidence in acute hemiplegia. NeuroRehabilitation. 2020;46(4):577-587. doi: 10.3233/NRE-203086. PMID 32538882
- [Background] Ronsse R, Puttemans V, Coxon JP, Goble DJ, Wagemans J, Wenderoth N, Swinnen SP. Motor learning with augmented feedback: modality-dependent behavioral and neural consequences. Cereb Cortex. 2011 Jun;21(6):1283-94. doi: 10.1093/cercor/bhq209. Epub 2010 Oct 28. PMID 21030486
- [Background] Rose DK, DeMark L, Fox EJ, Clark DJ, Wludyka P. A Backward Walking Training Program to Improve Balance and Mobility in Acute Stroke: A Pilot Randomized Controlled Trial. J Neurol Phys Ther. 2018 Jan;42(1):12-21. doi: 10.1097/NPT.0000000000000210. PMID 29232308
- [Background] Spencer J, Wolf SL, Kesar TM. Biofeedback for Post-stroke Gait Retraining: A Review of Current Evidence and Future Research Directions in the Context of Emerging Technologies. Front Neurol. 2021 Mar 30;12:637199. doi: 10.3389/fneur.2021.637199. eCollection 2021. PMID 33859607
- [Background] Steuer I, Guertin PA. Central pattern generators in the brainstem and spinal cord: an overview of basic principles, similarities and differences. Rev Neurosci. 2019 Jan 28;30(2):107-164. doi: 10.1515/revneuro-2017-0102. PMID 30543520